CLINICAL TRIAL: NCT05173649
Title: Effect of Calisthenics and Neuromuscular Training in Patients With Knee Osteoarthritis.
Brief Title: Calisthenic and Neuromuscular Training in Patients With Knee OA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00956 Tayyeba Majid
Record Dates: First submitted 2021-11-18; First posted 2021-12-30 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
Keywords: Calisthenic training; Neuromuscular training; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither subjects nor the investigator who is assessing the patient are aware of the treatment assignment until the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calisthenic Training (Experimental): Calisthenic Training Group
  Interventions: Other: Calisthenic Training; Other: Neuromuscular Training
- Neuromuscular Training Group (Experimental): Neuromuscular Training Group
  Interventions: Other: Calisthenic Training; Other: Neuromuscular Training

INTERVENTIONS:
Other: Calisthenic Training — Calisthenic Training Performed thrice a week after baseline assessment Standard Physical therapy treatment along with following exercises.
  1. Abductor-Adductor leg raise
  2. Alternate toe touch
  3. Knee Bend
  4. Prone leg extension
  5. Forward Lunges
  6. Toe Raise/ Calf raise Progressive training include following exercises.
  1. Leg Lifts 2. Jack Twists 3. Side Lunges 4. Short bridge 5. Calf Raise with weight.
  Other Names: Group A
Other: Neuromuscular Training — Neuromuscular Training Performed thrice a week after baseline assessment Standard Physical therapy treatment along with following exercises.
  1. Up and down step exercise in posterior and lateral directions.
  2. Walking in anterior and posterior
  3. Directions with eyes opened and eyes closed.
  4. Walking in lateral direction with eyes opened and eyes closed.
  5. Standing on one extremity
  6. Inclination in anterior and lateral direction with eyes opened and closed. Progressive training includes following exercises.
  1. Up and down on Bosu exercise. 2. Plantar flexion on minitrampoline. 3. Standing on one extremity on Bosu. 4. Standing on one extremity on minitrampoline
  Other Names: Group B

SUMMARY:
The aim of the study is to compare effects of calisthenics and neuromuscular training in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
OsteoArthristis (OA) is the most frequent form of arthritis and a leading cause of pain and disability worldwide. OA can affect any synovial joint, although the hip, knee, hand, foot and spine are the most commonly affected sites.

The knee is the most commonly affected joint and knee OA (KOA) represents the leading joint disorder in the world. At present, there is no preventive or curative drug treatment available for KOA.

Physical therapy plays a significant role in treating patients with knee OA. Rehabilitation enables the patient to cope with their daily task independently and mainly focus on self-help and patient-driven treatments rather than on passive therapies delivered by clinicians.

A systemic review was conducted on Comparative Effect of Calisthenics and Proprioceptive Exercises on Pain, Proprioception, Balance and Function in Chronic Osteoarthritis of Knee. According to this study Light intensity Calisthenics exercises are effective and can be recommended as an adjunct to conventional physiotherapy for the patients with Osteoarthritis knee.

Another research was conducted on Efficacy of Neuromuscular Training on Pain, Balance and Function in Patients with Grade I and II Knee Osteoarthritis. The results shows that although conventional exercise program is effective in reducing knee pain, and increasing lower extremity muscle strength and range of motion, adding neuromuscular training (KBA) along with conventional exercise program in rehabilitation leads to higher improvement on balance and function in patient with knee grade I and II osteoarthritis.

A positive effect has been observed in treating patients with both the interventions.

The past research records are evident that therapists have determined individual effects of calisthenics and neuromuscular training for rehabilitation of Knee OA. The evidence for implementation of two protocols for rehabilitation of Knee OA is sparse. So the aim of the study is to compare effects of calisthenics and neuromuscular training in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with chronic OA (symptoms for more than 3 months).
2. Subjects willing to participate and take treatment.
3. Grade of 2 to 3 as per Kellegren and Lawrence radiographic classification.

Exclusion Criteria:

1. Subjects having any systemic joint pathologies, inflammatory joint disease (e.g.

   Rheumatoid arthritis, gouty arthritis, psoriatic arthritis).
2. Subjects who had any neurological deficit (paresthesia, sensory loss, radiculopathy, myelopathy any mental illness (Dementia, Alzheimer's, Parkinson disease etc.) that can affect orientation and concentration.
3. Subjects on medication like antidepressants, corticosteroid, and anti-inflammatory medications.
4. Peripheral vascular diseases.
5. Any history of surgery related to lower extremity.
6. Subjects having metal implants in the lower limb

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) | 6 weeks
  Changes are measured from baseline. This test is used to measure physical function. The maximum score is 96 Higher the score the worst is pain, stiffness and physical function.
NPRS(Numeric pain rating scale) | 6 weeks
  Changes are measured from baseline. The test is used to measure pain. It score ranges from 0 to 10 with 0 indicating no pain and 10 is for pain as severe as possible
Short Physical Performance Battery | 6 weeks
  Changes are measured from baseline. The test is used to measure balance ,lower extremity strength and functional capacity with maximum score of 12. Score less than 10 indicates disability.
Mini BES-Test | 6 weeks
  Changes are measured from baseline. It is 36 items scales that evaluates Balance with total score of 28

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No